CLINICAL TRIAL: NCT05135494
Title: Effects of Inspiratory Muscle Training on the Severity of Obstructive Sleep Apnea in Individuals After Stroke: a Randomized and Controlled Clinical Trial
Brief Title: Effects of Inspiratory Muscle Training on the Severity of Obstructive Sleep Apnea in Individuals After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Network of Rehabilitation Hospitals (Other)
Responsible Party: Principal Investigator, Lorena de Oliveira Vaz Miranda, Principal Investigatot, Sarah Network of Rehabilitation Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 47173121.0.0000.0022
Record Dates: First submitted 2021-11-10; First posted 2021-11-26 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Obstructive Sleep Apnea; Inspiratory Muscle Training
MeSH Terms: conditions — Stroke; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group: Inspiratory Muscle Training + rehabilitation program
  Interventions: Other: Inspiratory Muscle Training
- Control Group (Other): Control Group: rehabilitation program
  Interventions: Other: Control

INTERVENTIONS:
Other: Inspiratory Muscle Training — The Experimental Group will perform IMT which includes training of the inspiratory muscles with the PowerBreath Medic Plus regulated at 75% of the subjects' maximal inspiratory pressure (MIP) values, five times/week over five weeks 5 sets of 5 repetitions with 1 set increasing each week.
  They will participate of the rehabilitation program that will consist of an average of 8 weekly sessions of physiotherapy and speech therapy, totaling 40 sessions. They will also perform 150 to 180 minutes of aerobic exercise of their choice and guidance on behavioral measures to manage OSA.
  Arms: Experimental Group
Other: Control — The control group will participate of the rehabilitation program that will consist of an average of 8 weekly sessions of physiotherapy and speech therapy, totaling 40 sessions. They will also perform 150 to 180 minutes of aerobic exercise of their choice and guidance on behavioral measures to manage OSA.
  Arms: Control Group

SUMMARY:
The prevalence of Obstructive Sleep Apnea (OSA) is high in individuals after a stroke. There are few studies evaluating the effects of inspiratory muscle training (IMT) in individuals with OSA and the findings regarding the possible effect on Apneia/Hipopneia Index (AHI) reduction are still controversial.

This study will test the hypothesis that training of the inspiratory muscles is effective in improving severity of OSA, sleep quality and daytime sleepiness in individuals after stroke participating in a rehabilitation program.

Methods: For this prospective, sigle blinded, randomized clinical trial, people after stroke will be randomly allocated into either experimental or control groups. The experimental group will undertake training of the inspiratory muscles with the PowerBreath Medic Plus regulated at 75% of the subjects' maximal inspiratory pressure (MIP) values, five times/week over five weeks 5 sets of 5 repetitions with 1 set increasing each week. Both groups will participate in the rehabilitation program and will receive the same dose of physiotherapy, speech therapy and aerobic exercise sessions. At baseline and post intervention after the cessation of the interventions, researchers blinded to group allocations will collect all outcome measures.

Study outcomes: Primary outcome will be OSA severity measured using the Apnea/Hypopnea Index (AHI). Secondary outcomes will include inspiratory endurance and pressure, functional independence, sleep quality and daytime sleepiness

DETAILED DESCRIPTION:
The prevalence of Obstructive Sleep Apnea (OSA) is high in individuals after a stroke. The gold standard treatment for OSA is the use of Positive Airway Pressure, but due to the low adherence to this resource, the multidisciplinary approach for the treatment of OSA is becoming the best therapeutic option. There are few studies evaluating the effects of inspiratory muscle training (IMT) in individuals with OSA and the findings regarding the possible effect on Apneia/Hipopneia Index (AHI) reduction are still controversial.

Aims:The primary objective of this study is to identify the effects of IMT on the severity of OSA in indivuals after stroke participating in a rehabilitation program. The secondary objectives are to identify effects of IMT on sleep quality and daytime sleepiness and analyze the correlation between severity of OSA and functional independence, inspiratory endurance and pressure.

Methods: For this prospective, sigle blinded, randomized clinical trial, people after stroke will be randomly allocated into either experimental or control groups. The experimental group will undertake training of the inspiratory muscles with the PowerBreath Medic Plus regulated at 75% of the subjects' maximal inspiratory pressure (MIP) values, five times/week over five weeks 5 sets of 5 repetitions with 1 set increasing each week. Both groups will participate in the rehabilitation program and will receive the same dose of physiotherapy, speech therapy and aerobic exercise sessions. At baseline and post intervention after the cessation of the interventions, researchers blinded to group allocations will collect all outcome measures.

Study outcomes: Primary outcome will be OSA severity measured using the Apnea/Hypopnea Index (AHI). Secondary outcomes will include inspiratory endurance and pressure, functional independence, sleep quality and daytime sleepiness

ELIGIBILITY:
Inclusion Criteria:

* Individuals after stroke of any etiology (ischemic or hemorrhagic), 18 to 80 years age, in a subacute or chronic phase (over 3 months to 5 years); with a diagnosis of OSA, defined as increased AHI (>5/h) in a polysomnography exam.

Exclusion Criteria:

* Individuals with BMI > 40, using Positive Airway Pressure during sleep, severe OSA (AHI > 30), previous diagnosis of severe nasal obstructive disease; craniofacial malformations including signs of dentoskeletal deformities, history of pharyngeal surgery to treat apnea, palatine tonsil hypertrophy (grade III and IV); edentulous people or users of complete dental prostheses; presence of oral apraxia; facial paralysis that prevents lip occlusion; aphasia that compromises the understanding of verbal commands; smokers and former smokers with less than 6 months of smoking cessation, orthopedic changes that include distortions of the rib cage and lung parenchyma diseases and that present other associated neurological diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
OSA severity | 5 weeks (immediately post intervention)
  OSA severity measured using the Apnea/Hypopnea Index (AHI)

SECONDARY OUTCOMES:
inspiratory muscle endurance | 5 weeks (immediately post intervention)
  inspiratory muscle endurance measured through the incremental endurance test
inspiratory muscular strength | 5 weeks (immediately post intervention)
  inspiratory muscular strength measured through inspiratory pressures
sleep quality | 1 month post intervention
  sleep quality measered through Pittisburgh Sleep Quality Index
daytime sleepiness | 1 month post intervention
  daytime sleepiness measered through Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Lorena de Oliveira Vaz, Salvador, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Oliveira Vaz L, Galvao AP, Nunes DLM, de Almeida JC, de Fatima Garcia Diniz J, Oliveira-Filho J. Effects of inspiratory muscle training on the severity of obstructive sleep apnea in individuals after stroke: a protocol for a randomized controlled trial. Sleep Breath. 2023 Dec;27(6):2257-2263. doi: 10.1007/s11325-023-02825-0. Epub 2023 Apr 27. PMID 37103682